CLINICAL TRIAL: NCT04090411
Title: A Phase 2B, Multicenter, Randomized, Double-Blind, Placebo-Controlled Dose-Ranging Study to Evaluate The Efficacy, Safety, and Pharmacokinetics of PF-06480605 in Adult Participants With Moderate To Severe Ulcerative Colitis
Brief Title: A Study to Evaluate the Efficacy and Safety of PF-06480605 in Adults With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XA45397; TL1A (Other: Alias Study Number); Tuscany 2 (Other: Alias Study Number); 2019-002698-74 (EudraCT Number); B7541007 (Other: Previous Study ID)
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Moderate to Severe Ulcerative Colitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Experimental): Induction - Placebo SC Q4W, (sub-cutaneous every 4 weeks) Chronic- PF-06480605 50 mg SC Q4W
  Interventions: Other: Induction- Placebo SC Q4W; Drug: Chronic- PF-06480605 50 mg SC Q4W
- Cohort 2 (Experimental): Induction - Placebo SC Q4W, Chronic- PF-06480605 150 mg SC Q4W
  Interventions: Other: Induction- Placebo SC Q4W; Drug: Chronic- PF-06480605 150 mg SC Q4W
- Cohort 3 (Experimental): Induction - Placebo SC Q4W, Chronic- PF-06480605 450 mg SC Q4W
  Interventions: Other: Induction- Placebo SC Q4W; Drug: Chronic- PF-06480605 450 mg SC Q4W
- Cohort 4 (Placebo Comparator): Induction- PF-06480605 50 mg SC Q4W, Chronic- PF-06480605 50 mg SC Q4W
  Interventions: Drug: Induction- PF-06480605 50 mg SC Q4W; Drug: Chronic- PF-06480605 50 mg SC Q4W
- Cohort 5 (Experimental): Induction- PF-06480605 150 mg SC Q4W, Chronic- PF-06480605 50 mg SC Q4W
  Interventions: Drug: Induction- PF-06480605 150 mg SC Q4W; Drug: Chronic- PF-06480605 50 mg SC Q4W
- Cohort 6 (Experimental): Induction- PF-06480605 150 mg SC Q4W, Chronic- PF-06480605 150 mg SC Q4W
  Interventions: Drug: Induction- PF-06480605 150 mg SC Q4W; Drug: Chronic- PF-06480605 150 mg SC Q4W
- Cohort 7 (Experimental): Induction- PF-06480605 450 mg SC Q4W, Chronic- PF-06480605 50 mg SC Q4W
  Interventions: Drug: Induction- PF-06480605 450 mg SC Q4W; Drug: Chronic- PF-06480605 50 mg SC Q4W
- Cohort 8 (Experimental): Induction- PF-06480605 450 mg SC Q4W, Chronic- PF-06480605 150 mg SC Q4W
  Interventions: Drug: Induction- PF-06480605 450 mg SC Q4W; Drug: Chronic- PF-06480605 150 mg SC Q4W
- Cohort 9 (Experimental): Induction- PF-06480605 450 mg SC Q4W, Chronic- PF-06480605 450 mg SC Q4W
  Interventions: Drug: Induction- PF-06480605 450 mg SC Q4W; Drug: Chronic- PF-06480605 450 mg SC Q4W

INTERVENTIONS:
Drug: Induction- PF-06480605 50 mg SC Q4W — PF-06480605
  Arms: Cohort 4
Drug: Induction- PF-06480605 150 mg SC Q4W — PF-06480605
  Arms: Cohort 5; Cohort 6
Drug: Induction- PF-06480605 450 mg SC Q4W — PF-06480605
  Arms: Cohort 7; Cohort 8; Cohort 9
Other: Induction- Placebo SC Q4W — 0 mg Placebo
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: Chronic- PF-06480605 50 mg SC Q4W — PF-06480605
  Arms: Cohort 1; Cohort 4; Cohort 5; Cohort 7
Drug: Chronic- PF-06480605 150 mg SC Q4W — PF-06480605
  Arms: Cohort 2; Cohort 6; Cohort 8
Drug: Chronic- PF-06480605 450 mg SC Q4W — PF-06480605
  Arms: Cohort 3; Cohort 9

SUMMARY:
This phase 2b study is designed to have all subjects go into a 12 week induction period to compare different doses of study drug against placebo. After induction is complete all subjects will receive active therapy for 40 weeks, followed by a 12 week follow up period.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of UC for >=3 months.
* Participants with moderate to severe active UC as defined by a Total Mayo Score of >=6, and an endoscopic subscore of >=2.
* Active disease beyond the rectum (>15 cm of active disease from the anal verge at the screening endoscopy).
* Must have failed or been intolerant to at least one of the following class of medications: steroids, immunosuppressants, anti-TNFs, anti-integrin inhibitors, anti- IL-12/23 inhibitors, or JAK inhibitors.

Exclusion Criteria:

* Participants with a diagnosis of ischemic colitis, infectious colitis, radiation colitis, microscopic colitis, indeterminate colitis, or findings suggestive of Crohn's disease (eg, skip lesions, fistulae/perianal disease, non-necrotizing granulomas, etc.).
* Participants with an imminent need for surgery or with elective surgery scheduled to occur during the study
* Chest Radiograph showing abnormalities: The study will accept a Chest x-ray or computed tomography scan of the chest examination performed up to 12 weeks prior to screening if available.
* 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results
* Infected with tuberculosis, (TB): Any evidence of untreated latent or active TB infection.
* Infected with human immunodeficiency virus, (HIV), Hepatitis B or C viruses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (164):
- United States (53):
  - Digestive Health Specialists, Dothan, Alabama
  - Dothan Surgery Center, Dothan, Alabama
  - Flowers Hospital, Dothan, Alabama
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Surinder Saini, M.D., Inc., Newport Beach, California
  - Endoscopy Center of Connecticut, LLC, Guilford, Connecticut
  - Endoscopy Center of Connecticut, LLC, Hamden, Connecticut
  - Medical Research Center Of Connecticut, LLC, Hamden, Connecticut
  - PACT Gastroenterology Center, Hamden, Connecticut
  - Whitney Imaging, Hamden, Connecticut
  - Medycal Research Inc., Brooksville, Florida
  - Safety Harbor Surgery, Clearwater, Florida
  - Trident Care, Clearwater, Florida
  - Tower Radiology Center, Oldsmar, Florida
  - Akumin, Tampa, Florida
  - Tampa Bay Endoscopy Center, Tampa, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - Gastroenterology Consultants P.C., Roswell, Georgia
  - The University of Chicago Medical Center (clinic address), Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital - Office, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Endoscopy Center, Farmington Hills, Michigan
  - Valley View Surgery Center, Las Vegas, Nevada
  - Sierra Clinical Research, Las Vegas, Nevada
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College, New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medical Center, New York, New York
  - Weill Cornell Medical College- New York Presbyterian Hospital, New York, New York
  - Investigational Drug Services, Philadelphia, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Gastroenterology Associates, PA of Greenville, Greenville, South Carolina
  - Vanderbilt GI Endoscopy Lab at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt Heart One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt Inflammatory Bowel Disease Clinic, Nashville, Tennessee
  - Vanderbilt Laboratory Services North One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt One Hundred Oaks Imaging, Nashville, Tennessee
  - Vanderbilt University Medical Center - GI Research Office, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Vanderbilt University Med. Center, Nashville, Tennessee
  - Vanderbilt University Medical Center- Heart Station (ECG), Nashville, Tennessee
  - PrimeCare Medical Group, Houston, Texas
  - Gastroenterology Consultants of San Antonio, PA, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - South Texas Radiology Imaging Centers, San Antonio, Texas
  - Gastroenterology Associates of Northern VA, Fairfax, Virginia
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia
  - Verity Research, Inc., Fairfax, Virginia
  - Medical Diagnostic Imaging, Wauwatosa, Wisconsin
  - Allegiance Internal Medicine and Allegiance Research Specialists, Wauwatosa, Wisconsin
  - GI Associates, Wauwatosa, Wisconsin
- Australia (3):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Mater Misericordiae Ltd., South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- University Hospitals Leuven/Department of Gastroenterology, Leuven, Belgium
- "ACIBADEM City Clinic Diagnostic-Consultative Center" EOOD, Sofia, Bulgaria
- Asociacion IPS Medicos Internistas de Caldas, Manizales, Caldas Department, Colombia
- France (7):
  - CHU d'Amiens-Picardie - SITE SUD, Amiens
  - Centre Hospitalier Regional Universitaire (CHU) de Lille - CIC, Lille
  - Centre Hospitalier Regional Universitaire (CHU) de Lille - Hopital Claude Huriez, Lille
  - Centre Hospitalier Regional Universitaire (CHU) de Lille, Lille
  - CHU Hôtel-Dieu, Nantes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Lyon Sud, Pierre-Bénite
- Germany (3):
  - Deutsches Rotes Kreuz Schwesternschaft Berlin Gemeinnützige Krankenhaus GmbH, Berlin
  - Studiengesellschaft BSF UG (haftungsbeschränkt), Halle
  - Studiengesellschaft BSF Unternehmergesellschaft, Halle
- Hungary (8):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred, Veszprém megye
  - Magyar Imre Kórház, Ajka
  - Clinexpert Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - Clinfan Kft., Szekszárd
  - Life Egészségcentrum, Székesfehérvár
  - Deák Jenő Kórház, Tapolca
  - Clinexpert Tatabanya, Szent Borbala Hospital, Tatabánya
  - Szofia Private Clinic, Veszprém
- India (7):
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Surat Institute of Digestive Sciences, Surat, Gujarat
  - Gujarat Hospital Gastro and Vascular Centre, Opp. Shree Ram Petrol Pump, Surat, Gujarat
  - M.S. Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - Grant Medical Foundation, Ruby Hall Clinic, Pune, Maharashtra
  - S.R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - S.M.S. Medical College & Hospital, Jaipur, Rajasthan
- Italy (6):
  - IRCCS "Saverio de Bellis", UOC Gastroenterologia, Castellana Grotte, BARI
  - Istituto Clinico Humanitas Centro per le Malattie Infiammatorie Croniche dell'Intestino - IBD Cent, Rozzano, Milan
  - A.O.U. dell'Università degli Studi della Campania "Luigi Vanvitelli", Napoli, Naples
  - Policlinico Universitario Campus Bio-Medico di Roma, Roma, RM
  - UO Malattie retto-Intestinali Ospedale "Sacro Cuore-don Calabria", Negrar, Verona
  - Azienda Ospedaliera di Padova - U.O.C. di Gastroenterologia, Padua
- Japan (8):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Tokyo Medical And Dental University Hospital, Bunkyo-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Fukuoka University Hospital, Fukuoka
- Mexico (4):
  - BRCR Global Mexico, Guadalajara, Jalisco
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion, Mérida, Yucatán
  - Karla Adriana Espinosa Bautista, Mexico City
  - Smiq S. de R.L. de C.V., Querétaro
- Poland (8):
  - KLIMED Marek Klimkiewicz, Bialystok
  - Indywidualna Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - MZ Badania Slowik Zymla Sp. j., Knurów
  - ENDOSKOPIA Sp. z o. o., Sopot
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - NZOZ Vivamed Jadwiga Miecz, Warsaw
  - Centrum Medyczne Melita Medical, Wroclaw
- Romania (2):
  - Medlife S.A., Bucharest
  - Spitalul Clinic Colentina, Bucharest
- Russia (12):
  - Pyatigorsk City Clinical Hospital, Pyatigorsk, Stavropol Kray
  - KDC "Evromedservis", OJSC, Moscow
  - Limited Liability Company "Medicinsky Center SibNovoMed", Novosibirsk
  - LLC Novosibirskiy Gastrocenter, Novosibirsk
  - Clinic of OSMU, Omsk
  - Perm Clinical Centre of the Federal Medical-Biological Agency, Perm
  - Private Healthcare Institution "Clinical Hospital" Russian Railways-Medicine "Samara city", Samara
  - Clinical Hospital named after S.R. Mirotvortsev, Saratov
  - Research Institute of Antimicrobial Chemotherapy, Smolensk
  - Tomsk Regional Clinical Hospital, Tomsk
  - City Hospital JSC "Medical centre", Tyumen
  - SBHI YaR "Regional Clinical Hospital", Yaroslavl
- Serbia (3):
  - Klinicki Centar Kragujevac, Kragujevac
  - Opsta Bolnica Subotica, Subotica
  - Opsta Bolnica "Djordje Joanovic", Odeljenje Interno, Odsek Gastroenterologija, Zrenjanin
- Slovakia (3):
  - KM Management spol. s.r.o., Nitra
  - Gastro LM s.r.o, Prešov
  - ENDOMED, s.r.o., Vranov nad Topľou
- South Africa (10):
  - Dr van Dyk & Partners Inc, Bloemfontein, Free State
  - IATROS International, Bloemfontein, Free State
  - Universitas Private Hospital, Bloemfontein, Free State
  - Ahmed Kathrada Private Hospital, Johannesburg, Gauteng
  - Lenasia Clinical Trial Centre, Johannesburg, Gauteng
  - Arwyp Medical Centre, Kempton Park, Gauteng
  - Clinresco Centres (Pty) Ltd, Kempton Park, Gauteng
  - Emmed Research, Pretoria, Gauteng
  - Radiology24 Jakaranda Hospital, Pretoria, Gauteng
  - Mediclinic Kloof Hospital, Pretoria, Gauteng
- Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid, Spain
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Faculty of Medicine, Chulalongkorn University, Pathum Wan, Bangkok
  - Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Phramongkutklao Hospital, Bangkok
- Turkey (Türkiye) (5):
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Kocaeli Universitesi Tip Fakultesi, Ic Hastaliklari Anabilim Dali, Kocaeli
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin
  - Bulent Ecevit Universitesi Tip Fakultesi, Zonguldak
- Ukraine (8):
  - Municipal non-profit enterprise of Kharkiv regional council "Regional clinical hospital", Kharkiv
  - Municipal non-profit enterprise "City clinical hospital #2 named after O.O.Shalimov", Kharkiv
  - Medical Centre Medical Clinic Blagomed LLC, Kyiv
  - Municipal Non-profit Enterprise "Kyiv City Clinical Hospital #1", Kyiv
  - Municipal Non-profit enterprise of Kyiv Regional Council "Kyiv regional hospital", Kyiv
  - Municipal non-profit enterprise of Kyiv regional council "Kyiv regional clinical hospital", Kyiv
  - Medical center of Limited Liability Company "Health Clinic", medical clinical research center, Vinnytsia
  - Medical Centre "DIACENTER" LLC, Zaporizhzhia
- United Kingdom (7):
  - Endoscopy Facility - Spire Little Aston Hospital, Sutton Coldfield, Birmingham
  - MeDiNova North London Quality Research Site, Northwood, Middlesex
  - MeDiNova Northamptonshire Quality Research Site, Corby
  - Egin Research Ltd, High Wycombe
  - Chest X-ray Facility - BMI Bishops Wood Hospital, Northwood
  - Spire Nottingham Hospital, Nottingham
  - Endoscopy Facility - Orpington Endoscopy Centre, Orpington

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Danese S, Allegretti JR, Schreiber S, Peyrin-Biroulet L, Jairath V, D'Haens G, Kierkus J, Leong RW, Yarur AJ, Vincent MS, Banerjee A, Chandra DE, Peeva E, Neelakantan S, Hung KE, McBride JM, Bojic D, Lasch K, Schiffman C, Feagan BG. Anti-TL1A antibody, afimkibart, in moderately-to-severely active ulcerative colitis (TUSCANY-2): a multicentre, double-blind, treat-through, multi-dose, randomised, placebo-controlled, phase 2b trial. Lancet Gastroenterol Hepatol. 2025 Oct;10(10):882-895. doi: 10.1016/S2468-1253(25)00129-3. Epub 2025 Jul 21. PMID 40706613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 246 participants with moderate to severe ulcerative colitis (UC) took part in the study at 114 investigative sites across 23 countries from 19 December 2019 to 25 October 2022. The study consisted of a 12-week induction period and a 40-week chronic therapy period.
Pre-assignment Details: Participants were randomized in 2:2:2:2:2:3:1:1:1 to 1 of 9 treatment sequences to receive PF-06480605 50 milligrams (mg), 150 mg, 450 mg or a matched placebo during the induction and chronic therapy periods. One participant in the PF-06480605 450 mg arm was enrolled but did not receive any treatment.
Groups:
- Induction Period: Placebo: Participants received PF-06480605 matching placebo, as a subcutaneous (SC) injection, every 4 weeks (Q4W) up to Week 12.
- Induction Period: PF-06480605 50 mg: Participants received PF-06480605, 50 mg, as a SC injection, Q4W up to Week 12.
- Induction Period: PF-06480605 150 mg: Participants received PF-06480605, 150 mg, as a SC injection, Q4W up to Week 12.
- Induction Period: PF-06480605 450 mg: Participants received PF-06480605, 450 mg, as a SC injection, Q4W up to Week 12.
- Placebo (Induction) to PF-06480605 (Chronic) 50 mg: Participants who received placebo and completed the 12-week induction period received PF-06480605, 50 mg, as a SC injection, Q4W from Week 16 to Week 52 in the chronic period.
- Placebo (Induction) to PF-06480605 (Chronic) 150 mg: Participants who received placebo and completed the 12-week induction period received PF-06480605, 150 mg, as a SC injection, Q4W from Week 16 to Week 52 in the chronic period.
- Placebo (Induction) to PF-06480605 (Chroinc) 450 mg: Participants who received placebo and completed the 12-week induction period received PF-06480605, 450 mg, as a SC injection, Q4W from Week 16 to Week 52 in the chronic period.
- PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg: Participants who received PF-06480605, 50 mg, and completed the 12-week induction period received PF-06480605, 50 mg, as a SC injection, Q4W from Week 16 to Week 52 in the chronic period.
- PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg: Participants who received PF-06480605, 150 mg, and completed the 12-week induction period received PF-06480605, 50 mg, as a SC injection, Q4W from Week 16 to Week 52 in the chronic period.
- PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg: Participants who received PF-06480605, 150 mg, and completed the 12-week induction period received PF-06480605, 150 mg, as a SC injection, Q4W from Week 16 to Week 52 in the chronic period.
- PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg: Participants who received PF-06480605, 450 mg, and completed the 12-week induction period received PF-06480605, 50 mg, as a SC injection, Q4W from Week 16 to Week 52 in the chronic period.
- PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg: Participants who received PF-06480605, 450 mg, and completed the 12-week induction period received PF-06480605, 150 mg, as a SC injection, Q4W from Week 16 to Week 52 in the chronic period.
- PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg: Participants who received PF-06480605, 450 mg, and completed the 12-week induction period received PF-06480605, 450 mg, as a SC injection, Q4W from Week 16 to Week 52 in the chronic period.
Period: Induction Period
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Started | 45 | 47 | 62 | 92 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 40 | 46 | 58 | 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 1 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Chronic Period
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Started | 0 | 0 | 0 | 0 | 12 | 14 | 14 | 46 | 27 | 30 | 26 | 26 | 29
Completed | 0 | 0 | 0 | 0 | 11 | 12 | 12 | 34 | 22 | 25 | 18 | 20 | 24
Not Completed | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 12 | 5 | 5 | 8 | 6 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 5 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 2 | 2 | 1 | 2
Not completed — Relocation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 3 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least one dose of investigational product (IP). Participants were analyzed according to the product they received.
Groups:
- Induction Period: Placebo: Participants received PF-06480605 matching placebo, as a SC injection, Q4W up to Week 12.
- Total: Total of all reporting groups
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg | Total
Number analyzed (Participants) | 45 | 47 | 62 | 91 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (12.90) | 37.8 (13.91) | 42.2 (13.02) | 41.6 (13.79) | 40.7 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 23 | 36 | 99
  Male | 24 | 28 | 39 | 55 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 3 | 10
  Not Hispanic or Latino | 42 | 43 | 55 | 86 | 226
  Unknown or Not Reported | 1 | 1 | 5 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 2 | 5
  Asian | 13 | 9 | 9 | 18 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 30 | 35 | 49 | 70 | 184
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 4 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Induction Period: Percentage of Participants Who Achieved Clinical Remission at Week 14
Description: Clinical remission was defined as total Mayo Score ≤2, with no individual subscore >1. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and physician's global assessment (PGA) subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease activity. Percentages have been rounded off to the nearest whole number.
Time Frame: At Week 14
Population: Evaluable population ITT included all participants randomly assigned to IP and who took at least one dose of IP in induction period. Participants were analyzed according to the product they received. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg
Number analyzed (Participants) | 43 | 47 | 60 | 88
percentage of participants | 11.6 [5.77 to 22.88] | 25.5 [15.44 to 37.19] | 23.3 [14.98 to 33.98] | 23.9 [16.58 to 32.06]
Statistical Analysis 1: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 50 mg; Test type: Superiority; p = 0.0545, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 13.90, 90% CI 2-sided [-0.20 to 27.65]
Statistical Analysis 2: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 150 mg; Test type: Superiority; p = 0.0823, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 11.71, 90% CI 2-sided [-1.70 to 24.09]
Statistical Analysis 3: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 450 mg; Test type: Superiority; p = 0.0642, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 12.24, 90% CI 2-sided [-0.64 to 22.91]

2. Primary Outcome: Induction Period: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs was defined as all events that started on or after the first dosing day and time, but before the last dose plus the lag time. An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. Results may differ from publications that used Week 14 as the end of the AE reporting timeframe.
Time Frame: From initiation of study treatment to either first dose in the chronic period or end of safety follow-up, whichever occurs first. (Approximately 16 weeks plus 12-week safety follow-up, if applicable.)
Population: Safety analysis population included all participants who received at least one dose of IP during the induction period. Participants were analyzed according to the product they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg
Number analyzed (Participants) | 45 | 47 | 62 | 91
Participants | 25 | 16 | 29 | 49

3. Primary Outcome: Induction Period: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. SAE was defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; or is a congenital anomaly/birth defect. Results may differ from publications that used Week 14 as the end of the AE reporting timeframe.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg
Number analyzed (Participants) | 45 | 47 | 62 | 91
Participants | 4 | 3 | 1 | 4

4. Primary Outcome: Induction Period: Number of Participants With AEs or SAEs Leading to Discontinuation
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. SAE was defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; or is a congenital anomaly/birth defect. Participants who had an AE/SAE that led to study discontinuation have been reported here. Results may differ from publications that used Week 14 as the end of the AE reporting timeframe.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg
Number analyzed (Participants) | 45 | 47 | 62 | 91
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Chronic Period: Number of Participants With TEAEs
Description: TEAEs was defined as all events that started on or after the first dosing day and time, but before the last dose plus the lag time. An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. Results may differ from publications that used Week 56 as the end of the AE reporting timeframe.
Time Frame: From first dose of study treatment in the chronic period to end of safety follow-up. (Approximately 40 weeks plus 12-week safety follow-up.)
Population: Evaluable population modified intent-to-treat (mITT) included all participants randomly assigned to IP who took at least one dose of IP in CPT. Participants were analyzed according to the treatment sequence they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 14 | 14 | 46 | 27 | 30 | 26 | 26 | 29
Participants | 5 | 9 | 9 | 30 | 16 | 15 | 18 | 18 | 20

6. Primary Outcome: Chronic Period: Number of Participants With SAEs
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. SAE was defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; or is a congenital anomaly/birth defect. Results may differ from publications that used Week 56 as the end of the AE reporting timeframe.
Time Frame: as for outcome 5
Population: Evaluable population mITT included all participants randomly assigned to IP who took at least one dose of IP in CPT. Participants were analyzed according to the treatment sequence they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 14 | 14 | 46 | 27 | 30 | 26 | 26 | 29
Participants | 0 | 0 | 0 | 5 | 1 | 0 | 2 | 1 | 4

7. Primary Outcome: Chronic Period: Number of Participants With AEs or SAEs Leading to Discontinuation
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. SAE was defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; or is a congenital anomaly/birth defect. Participants who had an AE/SAE that led to study discontinuation have been reported here. Results may differ from publications that used Week 56 as the end of the AE reporting timeframe.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 14 | 14 | 46 | 27 | 30 | 26 | 26 | 29
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Induction and Chronic: Percentage of Participants Who Achieved Remission as Per Food and Drug Administration (FDA) Definition 1 (Modified Remission 1)
Description: Modified remission 1 was defined as an endoscopic subscore = 0 (normal or inactive disease) or 1 (mild disease), stool frequency subscore = 0 (normal number of stools per day), and rectal bleeding subscore = 0 (no blood seen) at Week 14/Week 56. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and PGA subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease activity. Percentages have been rounded off to the nearest whole number.
Time Frame: Induction Period: At Week 14; Chronic Period: At Week 56
Population: Evaluable ITT and mITT populations included all participants randomly assigned to IP and who took at least one dose of IP in induction and chronic, respectively. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 43 | 47 | 60 | 88 | 12 | 13 | 14 | 42 | 27 | 26 | 25 | 24 | 28
percentage of participants | 7.0 [2.59 to 16.96] | 14.9 [8.05 to 25.12] | 13.3 [6.81 to 21.83] | 14.8 [9.50 to 21.77] | 16.7 [4.52 to 39.84] | 23.1 [8.80 to 46.97] | 21.4 [8.15 to 46.00] | 16.7 [9.06 to 27.68] | 22.2 [10.15 to 38.16] | 23.1 [10.56 to 39.84] | 16.0 [7.17 to 30.73] | 20.8 [10.50 to 36.99] | 17.9 [8.95 to 33.31]
Statistical Analysis 1: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 50 mg; Test type: Superiority; p = 0.1398, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 7.92, 90% CI 2-sided [-3.62 to 20.04]
Statistical Analysis 2: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 150 mg; Test type: Superiority; p = 0.2038, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 6.36, 90% CI 2-sided [-4.88 to 17.06]
Statistical Analysis 3: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 450 mg; Test type: Superiority; p = 0.1498, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 7.80, 90% CI 2-sided [-3.70 to 17.06]

9. Secondary Outcome: Induction and Chronic: Percentage of Participants Who Achieved Remission as Per FDA Definition 2 (Modified Remission 2)
Description: Modified remission 2 was defined as an endoscopic subscore = 0 (normal or inactive disease) or 1 (mild disease), ≥1 point decrease from baseline to achieve a stool frequency subscore = 0 (normal number of stools per day) or 1 (1 or 2 more stools than normal), and rectal bleeding subscore = 0 (no blood seen) at Week 14/Week 56. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and PGA subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease activity. Percentages have been rounded off to the nearest whole number.
Time Frame: Induction Period: At Week 14; Chronic Period: At Week 56
Population: as for outcome 8
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 43 | 47 | 60 | 88 | 12 | 13 | 14 | 42 | 27 | 26 | 25 | 24 | 28
percentage of participants | 11.6 [5.77 to 22.88] | 29.8 [19.94 to 42.34] | 35.0 [25.14 to 45.24] | 31.8 [23.65 to 40.77] | 50.0 [27.13 to 72.87] | 30.8 [14.16 to 54.45] | 35.7 [16.30 to 59.44] | 31.0 [19.38 to 43.33] | 33.3 [20.38 to 50.00] | 38.5 [23.32 to 56.43] | 28.0 [15.76 to 45.61] | 33.3 [17.80 to 52.14] | 35.7 [20.85 to 52.70]
Statistical Analysis 1: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 50 mg; Test type: Superiority; p = 0.0189, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 18.16, 90% CI 2-sided [3.25 to 32.23]
Statistical Analysis 2: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 150 mg; Test type: Superiority; p = 0.0045, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 23.37, 90% CI 2-sided [6.24 to 36.28]
Statistical Analysis 3: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 450 mg; Test type: Superiority; p = 0.0117, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 20.19, 90% CI 2-sided [3.22 to 31.31]

10. Secondary Outcome: Induction and Chronic: Percentage of Participants Who Achieved Endoscopic Improvement
Description: Endoscopic improvement was defined as an endoscopic subscore of 0 (Normal or inactive disease) or 1 (Mild disease [erythema, decreased vascular pattern, mild friability]) at Week 14/Week 56. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and PGA subscore. Each of the four assessments was rated with a score from 0 to 3. Higher scores indicate more severe disease activity. Percentages have been rounded off to the nearest whole number.
Time Frame: Induction Period: At Week 14; Chrnoic Period: At Week 56
Population: as for outcome 8
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 43 | 47 | 60 | 88 | 12 | 13 | 14 | 42 | 27 | 28 | 25 | 24 | 28
percentage of participants | 18.6 [9.61 to 30.24] | 40.4 [28.33 to 53.46] | 38.3 [27.81 to 48.61] | 40.9 [32.06 to 50.00] | 66.7 [39.84 to 84.58] | 38.5 [17.28 to 62.14] | 42.9 [22.38 to 64.51] | 38.1 [25.56 to 51.95] | 37.0 [22.12 to 54.66] | 39.3 [23.83 to 56.49] | 36.0 [21.43 to 54.39] | 37.5 [22.08 to 55.27] | 50.0 [33.31 to 66.69]
Statistical Analysis 1: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 50 mg; Test type: Superiority; p = 0.0146, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 21.82, 90% CI 2-sided [4.14 to 37.30]
Statistical Analysis 2: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 150 mg; Test type: Superiority; p = 0.0167, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 19.73, 90% CI 2-sided [2.76 to 34.05]
Statistical Analysis 3: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 450 mg; Test type: Superiority; p = 0.0094, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 22.30, 90% CI 2-sided [3.22 to 34.95]

11. Secondary Outcome: Induction and Chronic: Percentage of Participants Who Achieved Endoscopic Remission
Description: Endoscopic remission was defined as an endoscopic subscore of 0 (Normal or inactive disease) at Week 14/Week 56. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and PGA subscore. Each of the four assessments was rated with a score from 0 to 3. Higher scores indicate more severe disease activity. Percentages have been rounded off to the nearest whole number.
Time Frame: Induction Period: At Week 14; Chronic Period: At Week 56
Population: as for outcome 8
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 43 | 47 | 60 | 88 | 12 | 13 | 14 | 42 | 27 | 28 | 25 | 24 | 28
percentage of participants | 7.0 [2.59 to 16.96] | 19.1 [11.18 to 30.27] | 10.0 [4.45 to 18.01] | 10.2 [5.72 to 16.58] | 16.7 [4.52 to 39.84] | 23.1 [8.80 to 46.97] | 28.6 [13.09 to 54.00] | 11.9 [5.91 to 22.74] | 7.4 [1.99 to 20.38] | 7.1 [1.92 to 20.10] | 16.0 [7.17 to 30.73] | 8.3 [2.24 to 22.08] | 21.4 [9.77 to 36.62]
Statistical Analysis 1: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 50 mg; Test type: Superiority; p = 0.0489, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 12.17, 90% CI 2-sided [0.05 to 25.25]
Statistical Analysis 2: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 150 mg; Test type: Superiority; p = 0.3396, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 3.02, 90% CI 2-sided [-7.66 to 12.88]
Statistical Analysis 3: Comparison: Induction Period: Placebo vs Induction Period: PF-06480605 450 mg; Test type: Superiority; p = 0.3995, Chan and Zhang Method — One-sided P-value; Risk Difference (RD) = 3.25, 90% CI 2-sided [-7.42 to 11.58]

12. Secondary Outcome: Induction and Chronic: Trough Concentration (Ctrough) of PF-06480605
Time Frame: Induction Period: 30 mins postdose on Day 1, Weeks 4, 8, 12 and 14; Chronic Period: 30 mins postdose on Weeks 16, 20, 24, 28, 32, 36, 40, 44, 48; End of Treatment (EOT) (Week 52) and Follow-up (FU) Visits 1 (Week 56), 2 (Week 60) and 3 (Week 64)
Population: Pharmacokinetic (PK) population included all participants randomly assigned to IP and received at least one dose of PF-06480605 for whom at least one concentration value was reported. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 45 | 59 | 86 | 12 | 14 | 13 | 43 | 26 | 28 | 24 | 26 | 29
nanograms per milliliter (ng/mL)
  Postdose on Day 1: number analyzed (Participants) | 41 | 59 | 86 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Postdose on Day 1 | NA (NA) — The mean and standard deviation (SD) was not estimable as samples were below the limit of quantification (BLQ). | 1.227 (6.7722) | 1.279 (10.209) |  |  |  |  |  |  |  |  |
  Postdose on Week 4: number analyzed (Participants) | 45 | 58 | 85 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Postdose on Week 4 | 2251 (1122.5) | 6568 (3043.4) | 19660 (8637.7) |  |  |  |  |  |  |  |  |
  Postdose on Week 8: number analyzed (Participants) | 45 | 59 | 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Postdose on Week 8 | 2232 (1858.5) | 8381 (4769.8) | 25160 (12194) |  |  |  |  |  |  |  |  |
  Postdose on Week 12: number analyzed (Participants) | 45 | 55 | 82 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Postdose on Week 12 | 2181 (2080.3) | 8914 (5425.9) | 30900 (15724) |  |  |  |  |  |  |  |  |
  Postdose on Week 14: number analyzed (Participants) | 33 | 40 | 55 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Postdose on Week 14 | 4198 (3252.9) | 17110 (9380.6) | 49480 (18086) |  |  |  |  |  |  |  |  |
  Postdose on Week 16: number analyzed (Participants) | 0 | 0 | 0 | 11 | 13 | 13 | 42 | 24 | 28 | 24 | 25 | 29
  Postdose on Week 16 |  |  |  | NA (NA) — The mean and SD was not estimable as samples were BLQ. | 240.4 (862.23) | 6.123 (22.077) | 1969 (1932.7) | 9613 (6568.8) | 12450 (7605.4) | 39180 (19045) | 36320 (18215) | 32450 (17064)
  Postdose on Week 20: number analyzed (Participants) | 0 | 0 | 0 | 12 | 13 | 13 | 43 | 26 | 28 | 21 | 26 | 29
  Postdose on Week 20 |  |  |  | 2924 (1706.7) | 6680 (4188.0) | 25030 (9240.1) | 2516 (2279.8) | 5476 (4062.3) | 11500 (6289.0) | 19540 (10180) | 18200 (12244) | 34980 (17895)
  Postdose on Week 24: number analyzed (Participants) | 0 | 0 | 0 | 12 | 13 | 12 | 39 | 22 | 27 | 24 | 25 | 26
  Postdose on Week 24 |  |  |  | 2897 (1494.1) | 10990 (8884.5) | 29820 (15940) | 2956 (3018.7) | 4811 (3089.1) | 11090 (6765.1) | 10040 (6001.7) | 16890 (13735) | 35110 (16669)
  Postdose on Week 28: number analyzed (Participants) | 0 | 0 | 0 | 11 | 14 | 12 | 39 | 24 | 28 | 20 | 24 | 25
  Postdose on Week 28 |  |  |  | 2915 (2739.1) | 7587 (4748.7) | 38270 (12846) | 2613 (2763.5) | 3391 (2267.9) | 9840 (6630.1) | 5894 (3973.7) | 12920 (8418.9) | 35080 (14331)
  Postdose on Week 32: number analyzed (Participants) | 0 | 0 | 0 | 11 | 14 | 12 | 38 | 23 | 25 | 21 | 24 | 23
  Postdose on Week 32 |  |  |  | 2672 (2275.6) | 10520 (8027.4) | 38950 (21386) | 2330 (2253.4) | 3608 (3088.1) | 11790 (5931.7) | 5465 (3299.1) | 12060 (8871.1) | 36720 (16880)
  Postdose on Week 36: number analyzed (Participants) | 0 | 0 | 0 | 11 | 14 | 12 | 36 | 21 | 23 | 20 | 22 | 22
  Postdose on Week 36 |  |  |  | 3478 (2422.7) | 9279 (8345.1) | 36520 (20234) | 2802 (2573.3) | 3417 (2301.7) | 11680 (6728.9) | 4610 (2651.5) | 12360 (7217.1) | 33660 (14185)
  Postdose on Week 40: number analyzed (Participants) | 0 | 0 | 0 | 11 | 12 | 12 | 36 | 21 | 24 | 18 | 22 | 24
  Postdose on Week 40 |  |  |  | 2793 (1893.0) | 9246 (6289.2) | 41770 (18436) | 2820 (2590.1) | 3374 (2922.0) | 12050 (7678.1) | 3900 (2874.5) | 11830 (7571.4) | 33660 (11189)
  Postdose on Week 44: number analyzed (Participants) | 0 | 0 | 0 | 10 | 12 | 12 | 33 | 21 | 23 | 17 | 21 | 21
  Postdose on Week 44 |  |  |  | 3314 (2152.2) | 9346 (5199.5) | 45770 (20693) | 2867 (2655.4) | 3385 (3540.7) | 12190 (6504.8) | 3708 (2471.4) | 13060 (8745.9) | 36450 (12884)
  Postdose on Week 48: number analyzed (Participants) | 0 | 0 | 0 | 9 | 10 | 11 | 33 | 20 | 23 | 15 | 20 | 22
  Postdose on Week 48 |  |  |  | 2921 (2084.1) | 10750 (8216.0) | 46150 (19825) | 3159 (2810.1) | 3876 (3276.1) | 13230 (7740.3) | 4494 (3860.2) | 13700 (10253) | 38310 (13146)
  EOT (Week 52): number analyzed (Participants) | 0 | 0 | 0 | 10 | 9 | 12 | 28 | 21 | 19 | 17 | 19 | 24
  EOT (Week 52) |  |  |  | 3532 (2447.9) | 10510 (10337) | 49880 (21069) | 2848 (3037.0) | 3156 (2337.1) | 14580 (7988.8) | 4215 (3708.6) | 13930 (8673.4) | 40710 (15146)
  FU Visit 1 (Week 56): number analyzed (Participants) | 0 | 0 | 0 | 9 | 8 | 9 | 27 | 15 | 14 | 14 | 18 | 21
  FU Visit 1 (Week 56) |  |  |  | 4152 (3804.3) | 9755 (6903.0) | 43710 (26683) | 3246 (2965.2) | 3124 (2443.2) | 12870 (7884.4) | 4036 (3398.6) | 13410 (9499.7) | 43290 (17036)
  FU Visit 2 (Week 60): number analyzed (Participants) | 0 | 0 | 0 | 9 | 11 | 8 | 30 | 18 | 19 | 13 | 16 | 20
  FU Visit 2 (Week 60) |  |  |  | 1550 (1580.2) | 3797 (4065.6) | 19390 (13334) | 1092 (1232.9) | 1025 (858.32) | 4806 (2827.2) | 1285 (1436.1) | 5266 (5457.1) | 13930 (9036.0)
  FU Visit 3 (Week 64): number analyzed (Participants) | 0 | 0 | 0 | 8 | 11 | 8 | 29 | 17 | 19 | 17 | 17 | 17
  FU Visit 3 (Week 64) |  |  |  | 1099 (2081.3) | 1332 (2390.4) | 7976 (5279.5) | 766.1 (2372.9) | 257.3 (318.70) | 2011 (1752.1) | 825.8 (1883.2) | 1840 (2045.6) | 7136 (5642.6)

13. Secondary Outcome: Induction Period: Change From Baseline in Fecal Calprotectin
Time Frame: Baseline, Weeks 4, 8, and 12
Population: Biomarker analysis population included all participants randomly assigned to IP and who took at least one dose of PF-06480605 and in whom at least one measurement of biomarker of interest was reported. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per gram (µg/g)
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg
Number analyzed (Participants) | 37 | 41 | 55 | 82
micrograms per gram (µg/g)
  Baseline | 10.62 (2.145) | 9.99 (2.105) | 10.78 (2.120) | 10.23 (1.618)
  Change From Baseline at Week 4: number analyzed (Participants) | 35 | 36 | 49 | 79
  Change From Baseline at Week 4 | -0.32 (2.294) | -0.38 (1.973) | -1.24 (2.429) | -0.86 (2.618)
  Change From Baseline at Week 8: number analyzed (Participants) | 34 | 40 | 43 | 75
  Change From Baseline at Week 8 | -0.77 (2.601) | -1.28 (2.620) | -1.84 (2.779) | -1.69 (2.991)
  Change From Baseline at Week 12: number analyzed (Participants) | 34 | 35 | 44 | 74
  Change From Baseline at Week 12 | -0.62 (3.208) | -1.36 (2.837) | -2.43 (2.859) | -1.44 (3.003)

14. Secondary Outcome: Induction Period: Change From Baseline in High Sensitivity C-reactive Protein (hsCRP)
Time Frame: Baseline, Weeks 4, 8, and 12
Population: Biomarker analysis population included all participants randomly assigned to IP and who took at least one dose of PF-06480605 and in whom at least one measurement of biomarker of interest was reported. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg
Number analyzed (Participants) | 40 | 47 | 62 | 91
milligrams per deciliter (mg/dL)
  Baseline | 1.76 (2.135) | 1.47 (1.990) | 1.41 (1.799) | 1.82 (1.924)
  Change From Baseline at Week 4: number analyzed (Participants) | 40 | 46 | 61 | 89
  Change From Baseline at Week 4 | -0.49 (1.503) | -0.48 (1.669) | -0.75 (1.762) | -1.08 (1.577)
  Change From Baseline at Week 8: number analyzed (Participants) | 39 | 47 | 58 | 86
  Change From Baseline at Week 8 | -0.49 (1.929) | -0.45 (1.896) | -0.94 (2.120) | -1.09 (1.697)
  Change From Baseline at Week 12: number analyzed (Participants) | 38 | 43 | 54 | 82
  Change From Baseline at Week 12 | -0.96 (2.305) | -0.71 (1.764) | -1.25 (1.748) | -1.06 (1.834)

15. Secondary Outcome: Induction Period: Change From Baseline in Serum Soluble TL1A (sTL1A)
Time Frame: Baseline, Weeks 4, 8, and 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg
Number analyzed (Participants) | 39 | 42 | 58 | 88
picograms per milliliter (pg/mL)
  Baseline | 6.86 (0.441) | 6.74 (0.499) | 6.77 (0.534) | 6.83 (0.558)
  Change From Baseline at Week 4: number analyzed (Participants) | 39 | 40 | 56 | 86
  Change From Baseline at Week 4 | 0.01 (0.347) | 3.45 (1.097) | 3.85 (1.294) | 4.91 (0.834)
  Change From Baseline at Week 8: number analyzed (Participants) | 39 | 42 | 55 | 83
  Change From Baseline at Week 8 | -0.05 (0.549) | 3.14 (1.340) | 3.80 (1.486) | 4.88 (1.294)
  Change From Baseline at Week 12: number analyzed (Participants) | 36 | 40 | 53 | 81
  Change From Baseline at Week 12 | -0.02 (0.371) | 2.86 (1.666) | 3.72 (1.530) | 4.71 (1.908)

16. Secondary Outcome: Induction Period: Number of Participants With Anti-drug Antibodies (ADAs) and Neutralizing Antibodies (NAb) to PF-06480605
Description: Samples were considered to be positive for ADA against PF-06480605 if the titer was ≥ 60, and an ADA sample was considered to be negative if the titer was < 60. Samples were considered to be positive for NAb against PF-06480605 if the titer was ≥ 5, and an NAb sample was considered to be negative if the titer was < 5.
Time Frame: Baseline, Weeks 4, 8, 12, 14
Population: Evaluation of NAb is generally relevant only in participants who are positive for ADA. Immunogenicity analysis population included all participants randomly assigned to IP and who took at least one dose of PF-06480605 and in whom at least one post-treatment ADA determination was reported. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg
Number analyzed (Participants) | 45 | 59 | 88
Participants
  ADA at Baseline: number analyzed (Participants) | 41 | 59 | 88
  ADA at Baseline | 0 | 1 | 2
  NAb at Baseline: number analyzed (Participants) | 0 | 2 | 2
  NAb at Baseline |  | 0 | 0
  ADA at Week 4: number analyzed (Participants) | 45 | 58 | 86
  ADA at Week 4 | 29 | 16 | 24
  NAb at Week 4: number analyzed (Participants) | 33 | 27 | 35
  NAb at Week 4 | 1 | 0 | 0
  ADA at Week 8: number analyzed (Participants) | 45 | 58 | 84
  ADA at Week 8 | 39 | 34 | 34
  NAb at Week 8: number analyzed (Participants) | 44 | 41 | 41
  NAb at Week 8 | 10 | 4 | 1
  ADA at Week 12: number analyzed (Participants) | 44 | 56 | 82
  ADA at Week 12 | 41 | 36 | 36
  NAb at Week 12: number analyzed (Participants) | 42 | 40 | 46
  NAb at Week 12 | 12 | 7 | 3
  ADA at Week 14: number analyzed (Participants) | 45 | 54 | 83
  ADA at Week 14 | 41 | 35 | 33
  NAb at Week 14: number analyzed (Participants) | 42 | 39 | 38
  NAb at Week 14 | 14 | 7 | 3

17. Secondary Outcome: Chronic Period: Percentage of Participants Who Achieved Clinical Remission
Description: Clinical remission was defined as total Mayo Score ≤2, with no individual subscore >1. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and PGA subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease activity. Percentages have been rounded off to the nearest whole number.
Time Frame: At Week 56
Population: Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chronic period. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 13 | 14 | 42 | 27 | 26 | 25 | 24 | 28
percentage of participants | 33.3 [15.42 to 60.16] | 38.5 [17.28 to 62.14] | 35.7 [16.30 to 59.44] | 31.0 [19.38 to 43.33] | 29.6 [15.68 to 45.34] | 34.6 [20.86 to 52.62] | 24.0 [11.01 to 41.68] | 25.0 [11.49 to 42.28] | 39.3 [23.83 to 56.49]

18. Secondary Outcome: Chronic Period: Percentage of Participants Who Achieved Sustained Clinical Remission
Description: Clinical remission was defined as total Mayo Score ≤2, with no individual subscore >1. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and PGA subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease activity. Participants with sustained clinical remission were defined as those who achieved clinical remission at both Weeks 14 and 56. Percentages have been rounded off to the nearest whole number.
Time Frame: At Weeks 14 and 56
Population: Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chronic period. Overall number analyzed is the number of participants with data available for analysis. Participants were assessed at Week 56 if they achieved remission at Week 14. No participants in the Placebo (Induction) to PF-06480605 50 mg (Chronic) met the remission criteria at Week 14. Hence, this arm has been excluded.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 1 | 4 | 12 | 6 | 8 | 7 | 6 | 7
percentage of participants | 0 [0 to 0] | 25.0 [2.60 to 67.95] | 50.0 [27.13 to 72.87] | 50.0 [20.09 to 79.91] | 62.5 [28.92 to 85.31] | 28.6 [7.88 to 65.87] | 50.0 [20.09 to 79.91] | 85.7 [50.00 to 98.51]

19. Secondary Outcome: Chronic Period: Percentage of Participants Who Achieved Sustained Remission as Per FDA Definition 1 (Modified Remission 1)
Description: Modified remission 1 was defined as an endoscopic subscore = 0 (normal or inactive disease) or 1 (mild disease), stool frequency subscore = 0 (normal number of stools per day), and rectal bleeding subscore = 0 (no blood seen) at Week 14/Week 56. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and PGA subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease activity. Participants with sustained clinical remission were defined as those who achieved clinical remission at both Weeks 14 and 56. Percentages have been rounded off to the nearest whole number.
Time Frame: At Weeks 14 and 56
Population: Evaluable mITT population included all participants randomly assigned to IP and who took at least 1 dose of IP in the chronic period. Overall number analyzed is the number of participants with data available for analysis. Participants were assessed at Week 56 if they achieved remission at Week 14. No participants in Placebo (Induction) to PF-06480605 50 mg (Chronic) and Placebo (Induction) to PF-06480605 150 mg (Chronic) met remission criteria at Week 14. Hence, these arms have been excluded.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 3 | 7 | 5 | 3 | 4 | 3 | 5
percentage of participants | 33.3 [3.45 to 80.42] | 28.6 [7.88 to 65.87] | 40.0 [11.22 to 75.34] | 66.7 [19.58 to 96.55] | 25.0 [2.60 to 67.95] | 0 [0 to 53.58] | 80.0 [37.93 to 97.91]

20. Secondary Outcome: Chronic Period: Percentage of Participants Who Achieved Sustained Remission as Per FDA Definition 2 (Modified Remission 2)
Description: Modified remission 2 was defined as an endoscopic subscore = 0 (normal or inactive disease) or 1 (mild disease), ≥1 point decrease from baseline to achieve a stool frequency subscore = 0 (normal number of stools per day) or 1 = 1 or 2 more stools than normal, and rectal bleeding subscore = 0 (no blood seen) at Week 14/Week 56. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and PGA subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease activity. Participants with sustained clinical remission were defined as those who achieved clinical remission at both Weeks 14 and 56. Percentages have been rounded off to the nearest whole number.
Time Frame: At Weeks 14 and 56
Population: Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chronic period. Overall number analyzed is the number of participants with data available for analysis. Participants were assessed at Week 56 if they achieved remission at Week 14.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 1 | 1 | 3 | 14 | 10 | 11 | 9 | 10 | 8
percentage of participants | 0 [0.00 to 90.00] | 0 [0.00 to 90.00] | 33.3 [3.45 to 80.42] | 42.9 [22.38 to 64.51] | 70.0 [39.34 to 88.42] | 54.5 [30.24 to 80.04] | 33.3 [12.95 to 61.04] | 60.0 [34.08 to 81.24] | 75.0 [41.82 to 93.14]

21. Secondary Outcome: Chronic Period: Percentage of Participants Who Achieved Sustained Endoscopic Improvement
Description: Endoscopic improvement was defined as an endoscopic subscore of 0 (Normal or inactive disease) or 1 (Mild disease [erythema, decreased vascular pattern, mild friability]) at both Week 14 and Week 56. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and PGA subscore. Each of the four assessments was rated with a score from 0 to 3. Higher scores indicate more severe disease activity. Participants with sustained endoscopic improvement were defined as those who achieved improvement at both Weeks 14 and 56. Percentages have been rounded off to the nearest whole number.
Time Frame: At Weeks 14 and 56
Population: Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chronic period. Overall number analyzed is the number of participants with data available for analysis. Participants were assessed at Week 56 if they achieved improvement at Week 14.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 2 | 2 | 4 | 19 | 10 | 13 | 13 | 11 | 10
percentage of participants | 50.0 [5.13 to 94.87] | 0 [0.00 to 68.38] | 25.0 [2.60 to 67.95] | 47.4 [27.39 to 66.28] | 80.0 [50.00 to 94.55] | 61.5 [37.86 to 82.72] | 46.2 [24.55 to 71.30] | 63.6 [34.98 to 83.08] | 80.0 [50.00 to 94.55]

22. Secondary Outcome: Chronic Period: Percentage of Participants Who Achieved Sustained Endoscopic Remission
Description: Endoscopic remission was defined as an endoscopic subscore of 0 (Normal or inactive disease) at both Week 14 and Week 56. Mayo Score was a tool designed to measure disease activity for UC. The score ranges from 0 - 12 and was a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and PGA subscore. Each of the four assessments was rated with a score from 0 to 3. Higher scores indicate more severe disease activity. Participants with sustained endoscopic remission were defined as those who achieved endoscopic remission at both Weeks 14 and 56. Percentages have been rounded off to the nearest whole number.
Time Frame: At Weeks 14 and 56
Population: Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chronic period. Overall number analyzed is the number of participants with data available for analysis. Participants were assessed at Week 56 if they achieved remission at Week 14. No participants in Placebo (Induction) to PF-06480605 50 mg (Chronic) met remission criteria at Week 14. Hence, this arm has been excluded.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 2 | 1 | 9 | 2 | 4 | 3 | 2 | 3
percentage of participants | 0 [0.00 to 68.38] | 0 [0.00 to 90.00] | 22.2 [6.08 to 51.52] | 50.0 [5.13 to 94.87] | 25.0 [2.60 to 67.95] | 66.7 [19.58 to 96.55] | 50.0 [5.13 to 94.87] | 66.7 [19.58 to 96.55]

23. Secondary Outcome: Chronic Period: Change From Week 16 in Fecal Calprotectin
Time Frame: Week 16 (baseline), Weeks 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, and 64
Population: Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chronic period. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 11 | 12 | 43 | 23 | 27 | 22 | 24 | 29
μg/g
  Week 16 | 10.22 (1.414) | 9.28 (2.578) | 9.77 (2.347) | 8.86 (2.728) | 9.03 (2.765) | 7.72 (2.642) | 9.34 (2.500) | 8.39 (2.368) | 9.21 (2.438)
  Change From Week 16 at Week 20: number analyzed (Participants) | 12 | 10 | 12 | 39 | 23 | 27 | 21 | 23 | 29
  Change From Week 16 at Week 20 | -0.40 (1.174) | -1.46 (2.251) | -1.32 (1.956) | -0.31 (2.114) | 0.26 (2.247) | 0.43 (1.403) | -0.32 (1.740) | 0.18 (2.569) | -0.46 (1.435)
  Change From Week 16 at Week 24: number analyzed (Participants) | 12 | 10 | 12 | 41 | 21 | 26 | 19 | 24 | 28
  Change From Week 16 at Week 24 | -0.71 (1.302) | -0.84 (1.718) | -1.47 (3.331) | 0.24 (2.242) | -0.15 (2.433) | 0.36 (2.638) | -0.16 (1.874) | -0.30 (1.619) | 0.10 (1.892)
  Change From Week 16 at Week 28: number analyzed (Participants) | 12 | 11 | 11 | 37 | 21 | 24 | 20 | 22 | 23
  Change From Week 16 at Week 28 | -1.55 (1.984) | -1.17 (3.018) | -1.48 (1.817) | -0.16 (2.928) | -0.15 (2.409) | 0.03 (1.996) | -0.32 (2.440) | -0.16 (1.716) | -0.53 (2.136)
  Change From Week 16 at Week 32: number analyzed (Participants) | 10 | 11 | 11 | 36 | 21 | 20 | 19 | 21 | 24
  Change From Week 16 at Week 32 | -0.91 (2.497) | -1.36 (3.553) | -2.47 (3.044) | 0.21 (2.321) | -0.32 (2.516) | 0.31 (2.453) | -0.13 (2.192) | 0.17 (2.102) | -0.08 (1.491)
  Change From Week 16 at Week 36: number analyzed (Participants) | 11 | 10 | 11 | 32 | 19 | 21 | 17 | 22 | 21
  Change From Week 16 at Week 36 | -0.68 (2.353) | -1.83 (2.542) | -2.36 (4.202) | -0.37 (2.465) | -0.21 (2.584) | 0.50 (2.152) | -0.67 (1.889) | -0.36 (2.362) | -0.32 (1.724)
  Change From Week 16 at Week 40: number analyzed (Participants) | 11 | 10 | 11 | 34 | 17 | 21 | 15 | 19 | 24
  Change From Week 16 at Week 40 | -1.62 (1.814) | 0.22 (3.962) | -2.59 (2.493) | 0.17 (2.604) | 0.02 (1.779) | 0.35 (2.179) | 0.01 (2.696) | -0.42 (1.672) | -0.62 (2.434)
  Change From Week 16 at Week 44: number analyzed (Participants) | 11 | 9 | 11 | 32 | 19 | 20 | 14 | 18 | 22
  Change From Week 16 at Week 44 | -0.68 (2.015) | -1.48 (2.693) | -1.81 (2.705) | -0.09 (2.023) | -0.98 (2.089) | 0.02 (2.568) | 0.21 (2.377) | -0.97 (1.890) | -0.69 (1.737)
  Change From Week 16 at Week 48: number analyzed (Participants) | 11 | 10 | 11 | 31 | 19 | 20 | 14 | 19 | 24
  Change From Week 16 at Week 48 | -0.85 (1.843) | -1.01 (3.642) | -2.56 (3.178) | 0.60 (2.255) | -0.78 (2.542) | 0.09 (3.320) | 0.03 (3.027) | -0.54 (2.248) | -0.47 (2.150)
  Change From Week 16 at Week 52: number analyzed (Participants) | 11 | 10 | 11 | 32 | 17 | 19 | 13 | 15 | 23
  Change From Week 16 at Week 52 | -1.39 (1.922) | -0.39 (3.222) | -2.84 (2.668) | -0.02 (2.327) | -0.12 (1.386) | 0.09 (2.558) | -0.20 (3.294) | -0.61 (2.259) | -0.75 (2.355)
  Change From Week 16 at Week 60: number analyzed (Participants) | 10 | 7 | 9 | 28 | 16 | 15 | 11 | 14 | 20
  Change From Week 16 at Week 60 | -1.31 (2.119) | -0.09 (1.780) | -1.96 (3.041) | 0.36 (3.169) | -0.60 (1.840) | 0.17 (2.939) | 1.61 (1.426) | -0.91 (2.915) | -0.95 (2.131)
  Change From Week 16 at Week 64: number analyzed (Participants) | 10 | 8 | 9 | 27 | 16 | 16 | 12 | 15 | 20
  Change From Week 16 at Week 64 | -0.54 (2.208) | -1.48 (2.426) | -0.86 (2.562) | 0.58 (2.705) | 0.29 (1.834) | 0.10 (3.982) | 0.85 (3.321) | -1.18 (4.080) | -0.82 (2.007)

24. Secondary Outcome: Chronic Period: Change From Week 14 in hsCRP
Time Frame: Week 14 (baseline), Weeks 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 14 | 14 | 46 | 26 | 30 | 26 | 26 | 29
mg/dL
  Week 14 | 1.22 (1.667) | 2.49 (2.149) | 0.43 (2.484) | 0.72 (2.322) | 0.26 (1.898) | 0.11 (1.724) | 0.49 (2.152) | 0.56 (1.843) | 1.55 (1.376)
  Change From Week 14 at Week 16: number analyzed (Participants) | 12 | 12 | 13 | 45 | 25 | 30 | 25 | 25 | 29
  Change From Week 14 at Week 16 | -0.17 (0.745) | -0.32 (1.057) | -0.05 (1.622) | 0.12 (0.895) | 0.28 (1.218) | 0.04 (1.074) | -0.18 (1.247) | -0.21 (1.390) | -0.12 (1.283)
  Change From Week 14 at Week 20: number analyzed (Participants) | 12 | 14 | 14 | 42 | 25 | 29 | 25 | 25 | 29
  Change From Week 14 at Week 20 | -0.41 (1.420) | -1.06 (1.370) | -0.48 (2.403) | 0.34 (1.390) | 0.32 (1.449) | 0.48 (1.736) | -0.22 (1.141) | 0.68 (2.359) | -0.19 (1.362)
  Change From Week 14 at Week 24: number analyzed (Participants) | 12 | 14 | 14 | 42 | 23 | 28 | 24 | 26 | 27
  Change From Week 14 at Week 24 | -0.76 (1.232) | -1.52 (1.440) | -1.01 (2.445) | 0.28 (1.328) | 0.23 (1.063) | 0.06 (0.882) | -0.20 (1.391) | -0.13 (1.372) | -0.16 (1.387)
  Change From Week 14 at Week 28: number analyzed (Participants) | 11 | 13 | 12 | 39 | 22 | 28 | 22 | 24 | 26
  Change From Week 14 at Week 28 | -1.01 (1.398) | -1.12 (1.917) | -0.36 (1.665) | 0.31 (1.362) | 0.29 (1.156) | 0.26 (1.050) | -0.28 (1.546) | -0.25 (1.347) | -0.23 (1.044)
  Change From Week 14 at Week 32: number analyzed (Participants) | 11 | 14 | 13 | 40 | 24 | 25 | 23 | 24 | 24
  Change From Week 14 at Week 32 | -0.32 (1.893) | -0.79 (1.535) | -0.85 (2.253) | 0.30 (1.720) | 0.32 (1.565) | 0.72 (1.347) | -0.56 (1.572) | 0.28 (1.474) | -0.29 (1.347)
  Change From Week 14 at Week 36: number analyzed (Participants) | 11 | 14 | 13 | 36 | 22 | 25 | 21 | 24 | 22
  Change From Week 14 at Week 36 | -1.04 (2.335) | -1.29 (1.786) | -0.67 (2.760) | 0.07 (1.430) | 0.29 (1.490) | 0.28 (1.179) | -0.43 (1.507) | 0.36 (2.013) | -0.24 (1.614)
  Change From Week 14 at Week 40: number analyzed (Participants) | 11 | 13 | 12 | 33 | 20 | 25 | 19 | 23 | 23
  Change From Week 14 at Week 40 | -0.50 (1.893) | -1.09 (1.827) | -1.56 (2.351) | 0.17 (1.596) | 0.16 (1.432) | 0.31 (1.206) | -0.35 (1.645) | 0.19 (1.252) | -0.66 (1.154)
  Change From Week 14 at Week 44: number analyzed (Participants) | 11 | 12 | 12 | 34 | 21 | 22 | 18 | 22 | 22
  Change From Week 14 at Week 44 | -0.11 (1.709) | -1.31 (1.707) | -1.28 (2.448) | -0.06 (1.589) | -0.15 (1.612) | 0.66 (1.083) | 0.05 (1.513) | 0.20 (1.457) | -0.75 (1.272)
  Change From Week 14 at Week 48: number analyzed (Participants) | 10 | 12 | 12 | 33 | 21 | 23 | 18 | 21 | 23
  Change From Week 14 at Week 48 | -0.59 (1.596) | -1.29 (1.700) | -1.23 (2.619) | 0.28 (1.749) | 0.31 (1.314) | 0.21 (1.213) | 0.07 (0.985) | 0.07 (1.674) | -0.53 (1.254)
  Change From Week 14 at Week 52: number analyzed (Participants) | 11 | 12 | 12 | 33 | 21 | 23 | 19 | 20 | 22
  Change From Week 14 at Week 52 | -0.01 (2.228) | -1.05 (1.726) | -1.59 (2.195) | 0.10 (1.248) | 0.09 (1.299) | -0.13 (0.985) | 0.43 (1.144) | -0.02 (1.760) | -0.63 (1.221)
  Change From Week 14 at Week 56: number analyzed (Participants) | 10 | 10 | 10 | 29 | 19 | 21 | 16 | 19 | 22
  Change From Week 14 at Week 56 | -0.28 (1.346) | -0.92 (1.776) | -0.57 (1.766) | 0.25 (1.525) | 0.17 (1.998) | 0.21 (1.129) | 0.65 (0.994) | 0.31 (1.801) | -0.34 (1.463)
  Change From Week 14 at Week 60: number analyzed (Participants) | 9 | 11 | 10 | 30 | 20 | 20 | 16 | 17 | 21
  Change From Week 14 at Week 60 | -0.50 (2.114) | -0.93 (1.857) | -0.63 (2.397) | 0.40 (1.804) | 1.21 (1.844) | 0.51 (0.992) | 0.14 (1.395) | -0.55 (1.390) | -0.91 (1.643)
  Change From Week 14 at Week 64: number analyzed (Participants) | 10 | 11 | 10 | 28 | 21 | 22 | 17 | 17 | 17
  Change From Week 14 at Week 64 | 0.35 (1.750) | -0.97 (2.090) | -1.12 (2.366) | 0.28 (1.633) | 0.33 (1.848) | 0.22 (1.699) | 0.52 (1.659) | -0.06 (2.231) | -0.64 (1.802)

25. Secondary Outcome: Chronic Period: Change From Week 14 in Serum sTL1A
Time Frame: Week 14 (baseline), Weeks 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Population: Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chornic period. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 13 | 14 | 46 | 25 | 29 | 25 | 26 | 29
pg/mL
  Week 14 | 6.84 (0.443) | 7.21 (1.254) | 6.67 (0.463) | 9.78 (1.421) | 10.71 (1.543) | 10.61 (1.488) | 11.30 (2.495) | 11.34 (1.752) | 11.83 (0.726)
  Change From Week 14 at Week 16: number analyzed (Participants) | 11 | 12 | 13 | 44 | 23 | 27 | 25 | 25 | 29
  Change From Week 14 at Week 16 | -0.13 (0.576) | 0.29 (0.328) | 0.12 (0.330) | -0.03 (0.431) | -0.16 (0.302) | 0.03 (0.494) | 0.00 (0.987) | -0.26 (0.510) | -0.35 (0.435)
  Change From Week 14 at Week 20: number analyzed (Participants) | 12 | 13 | 13 | 44 | 25 | 27 | 23 | 26 | 29
  Change From Week 14 at Week 20 | 3.97 (0.722) | 3.43 (1.840) | 5.42 (0.954) | -0.03 (0.675) | -0.36 (0.645) | -0.01 (0.762) | -0.22 (1.086) | -0.74 (0.638) | -0.61 (0.780)
  Change From Week 14 at Week 24: number analyzed (Participants) | 12 | 12 | 13 | 41 | 21 | 26 | 23 | 25 | 27
  Change From Week 14 at Week 24 | 2.85 (1.141) | 3.84 (1.872) | 5.65 (0.909) | -0.02 (0.999) | -0.59 (0.912) | -0.41 (1.518) | -0.60 (1.133) | -0.90 (0.831) | -0.70 (1.047)
  Change From Week 14 at Week 28: number analyzed (Participants) | 12 | 13 | 12 | 39 | 23 | 27 | 22 | 24 | 26
  Change From Week 14 at Week 28 | 2.96 (1.033) | 3.78 (1.759) | 5.88 (0.731) | -0.16 (1.032) | -0.69 (1.036) | -0.33 (1.531) | -0.78 (1.384) | -0.87 (1.017) | -0.65 (1.047)
  Change From Week 14 at Week 32: number analyzed (Participants) | 11 | 13 | 13 | 40 | 22 | 25 | 22 | 24 | 24
  Change From Week 14 at Week 32 | 3.18 (1.346) | 3.65 (1.749) | 5.87 (0.588) | -0.10 (1.158) | -0.73 (1.092) | -0.07 (0.857) | -1.08 (1.337) | -0.93 (0.935) | -0.67 (0.914)
  Change From Week 14 at Week 36: number analyzed (Participants) | 10 | 13 | 13 | 36 | 22 | 24 | 20 | 22 | 23
  Change From Week 14 at Week 36 | 3.35 (1.185) | 3.53 (1.811) | 5.77 (0.745) | 0.06 (1.285) | -0.80 (1.036) | 0.01 (0.743) | -1.28 (1.630) | -0.81 (0.992) | -0.60 (0.812)
  Change From Week 14 at Week 40: number analyzed (Participants) | 11 | 12 | 12 | 35 | 20 | 25 | 18 | 23 | 24
  Change From Week 14 at Week 40 | 3.45 (0.990) | 3.17 (1.909) | 5.66 (0.926) | 0.04 (1.243) | -0.95 (1.188) | -0.01 (0.919) | -1.32 (1.739) | -0.75 (1.017) | -0.67 (0.891)
  Change From Week 14 at Week 44: number analyzed (Participants) | 11 | 11 | 12 | 36 | 21 | 24 | 18 | 22 | 24
  Change From Week 14 at Week 44 | 3.41 (1.068) | 3.09 (1.640) | 5.58 (1.106) | -0.01 (1.289) | -0.83 (1.282) | -0.11 (0.634) | -1.35 (1.812) | -0.60 (0.958) | -0.59 (0.873)
  Change From Week 14 at Week 48: number analyzed (Participants) | 11 | 11 | 12 | 34 | 21 | 24 | 17 | 21 | 23
  Change From Week 14 at Week 48 | 3.36 (1.108) | 2.83 (1.601) | 5.73 (1.029) | 0.03 (1.138) | -0.79 (1.198) | 0.14 (0.779) | -1.25 (1.554) | -0.54 (1.145) | -0.47 (0.853)
  Change From Week 14 at Week 52: number analyzed (Participants) | 11 | 11 | 12 | 33 | 21 | 23 | 18 | 20 | 25
  Change From Week 14 at Week 52 | 3.59 (1.128) | 2.83 (1.875) | 5.74 (1.224) | 0.06 (1.119) | -0.65 (1.090) | 0.26 (0.675) | -1.49 (1.711) | -0.54 (1.031) | -0.55 (1.134)
  Change From Week 14 at Week 56: number analyzed (Participants) | 10 | 11 | 10 | 30 | 18 | 22 | 16 | 19 | 23
  Change From Week 14 at Week 56 | 3.72 (1.114) | 2.71 (1.999) | 5.69 (1.173) | 0.31 (1.155) | -0.57 (1.191) | 0.26 (0.976) | -1.36 (1.870) | -0.29 (0.990) | -0.33 (0.919)
  Change From Week 14 at Week 60: number analyzed (Participants) | 9 | 10 | 10 | 32 | 20 | 20 | 15 | 16 | 22
  Change From Week 14 at Week 60 | 2.95 (1.646) | 2.87 (1.505) | 5.37 (1.556) | -0.08 (1.557) | -0.60 (1.303) | -0.13 (0.924) | -1.55 (1.985) | -0.70 (1.583) | -0.64 (0.929)
  Change From Week 14 at Week 64: number analyzed (Participants) | 10 | 10 | 9 | 29 | 21 | 21 | 15 | 18 | 21
  Change From Week 14 at Week 64 | 3.15 (1.775) | 2.88 (1.730) | 4.83 (1.860) | -0.28 (1.391) | -0.68 (1.200) | -0.19 (0.823) | -1.45 (2.361) | -0.97 (1.697) | -0.75 (1.062)

26. Secondary Outcome: Change From Baseline in Fecal Calprotectin Through the End of Study
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 60, and 64
Population: Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chronic period. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point. As pre-specified in the statistical analysis plan (SAP), data is presented using the treatment sequence in the chronic period.
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 11 | 14 | 40 | 27 | 26 | 23 | 21 | 28
μg/g
  Baseline: number analyzed (Participants) | 12 | 11 | 14 | 40 | 24 | 26 | 23 | 21 | 28
  Baseline | 10.43 (1.530) | 11.06 (1.450) | 10.44 (2.984) | 9.91 (2.069) | 11.12 (1.472) | 10.38 (2.683) | 10.41 (1.218) | 9.95 (2.225) | 10.23 (1.446)
  Change From Baseline at Week 4: number analyzed (Participants) | 12 | 11 | 12 | 36 | 22 | 23 | 22 | 20 | 28
  Change From Baseline at Week 4 | 0.41 (2.745) | -0.21 (0.925) | -1.15 (2.572) | -0.38 (1.973) | -1.56 (1.722) | -1.03 (3.037) | -1.28 (3.038) | -0.80 (2.727) | -0.69 (2.513)
  Change From Baseline at Week 8: number analyzed (Participants) | 10 | 10 | 14 | 39 | 20 | 21 | 22 | 20 | 28
  Change From Baseline at Week 8 | -0.36 (1.169) | -0.56 (1.601) | -1.21 (3.752) | -1.27 (2.652) | -2.03 (2.251) | -1.69 (3.357) | -2.29 (3.142) | -1.76 (3.108) | -1.27 (2.874)
  Change From Baseline at Week 12: number analyzed (Participants) | 11 | 9 | 14 | 35 | 18 | 24 | 21 | 21 | 28
  Change From Baseline at Week 12 | 0.46 (2.788) | -0.84 (2.026) | -1.32 (4.008) | -1.36 (2.837) | -2.62 (2.563) | -2.42 (3.174) | -1.21 (3.159) | -1.75 (3.477) | -1.31 (2.634)
  Change From Baseline at Week 16: number analyzed (Participants) | 12 | 10 | 12 | 37 | 21 | 25 | 21 | 20 | 28
  Change From Baseline at Week 16 | -0.21 (1.742) | -1.73 (2.941) | -0.67 (3.908) | -1.48 (3.378) | -2.30 (2.662) | -2.55 (2.883) | -0.87 (3.039) | -1.26 (3.043) | -1.08 (2.368)
  Change From Baseline at Week 20: number analyzed (Participants) | 12 | 10 | 14 | 39 | 23 | 25 | 22 | 19 | 28
  Change From Baseline at Week 20 | -0.61 (2.247) | -2.48 (2.935) | -2.35 (3.701) | -1.71 (3.104) | -1.87 (2.328) | -2.10 (2.824) | -1.61 (3.685) | -1.70 (3.353) | -1.55 (2.490)
  Change From Baseline at Week 24: number analyzed (Participants) | 12 | 10 | 14 | 38 | 22 | 24 | 19 | 21 | 27
  Change From Baseline at Week 24 | -0.92 (2.115) | -1.68 (2.505) | -2.52 (3.263) | -1.00 (3.050) | -2.31 (2.910) | -2.29 (3.768) | -1.25 (2.899) | -1.52 (3.478) | -0.95 (2.877)
  Change From Baseline at Week 28: number analyzed (Participants) | 12 | 11 | 12 | 32 | 21 | 22 | 21 | 18 | 22
  Change From Baseline at Week 28 | -1.76 (2.456) | -3.08 (3.021) | -2.70 (2.246) | -1.31 (3.225) | -2.46 (2.750) | -2.85 (3.782) | -1.60 (3.431) | -1.58 (3.213) | -1.61 (2.428)
  Change From Baseline at Week 32: number analyzed (Participants) | 10 | 11 | 12 | 35 | 27 | 20 | 20 | 17 | 24
  Change From Baseline at Week 32 | -1.43 (2.920) | -2.45 (2.916) | -2.87 (2.951) | -1.19 (3.384) | -2.62 (2.906) | -2.61 (3.609) | -1.56 (3.253) | -1.48 (3.014) | -1.31 (2.032)
  Change From Baseline at Week 36: number analyzed (Participants) | 11 | 10 | 12 | 30 | 21 | 21 | 17 | 18 | 20
  Change From Baseline at Week 36 | -1.05 (2.958) | -3.14 (2.233) | -3.11 (3.401) | -1.80 (3.019) | -2.39 (2.680) | -2.31 (3.468) | -2.11 (3.406) | -2.08 (3.070) | -2.05 (2.502)
  Change From Baseline at Week40: number analyzed (Participants) | 11 | 9 | 12 | 31 | 19 | 20 | 15 | 17 | 23
  Change From Baseline at Week40 | -1.99 (2.555) | -1.30 (2.745) | -3.02 (2.912) | -1.35 (3.354) | -2.17 (2.130) | -2.24 (3.311) | -1.58 (3.128) | -1.73 (3.158) | -1.87 (2.751)
  Change From Baseline at Week 44: number analyzed (Participants) | 11 | 8 | 12 | 31 | 21 | 20 | 14 | 15 | 21
  Change From Baseline at Week 44 | -1.05 (2.653) | -1.87 (2.871) | -2.35 (2.768) | -1.60 (3.435) | -2.93 (2.999) | -2.96 (3.311) | -1.09 (3.077) | -2.41 (3.338) | -2.08 (2.932)
  Change From Baseline at Week 48: number analyzed (Participants) | 11 | 9 | 12 | 29 | 21 | 19 | 14 | 16 | 23
  Change From Baseline at Week 48 | -1.22 (2.640) | -1.95 (3.001) | -2.87 (4.006) | -0.78 (2.906) | -2.81 (2.789) | -2.89 (3.346) | -1.74 (3.257) | -1.46 (3.800) | -1.75 (2.562)
  Change From Baseline at Week 52: number analyzed (Participants) | 11 | 9 | 12 | 30 | 20 | 17 | 13 | 12 | 22
  Change From Baseline at Week 52 | -1.76 (2.420) | -1.53 (2.796) | -3.27 (2.568) | -1.36 (3.019) | -2.20 (2.564) | -2.50 (3.129) | -1.90 (3.306) | -2.20 (2.991) | -2.07 (2.400)
  Change From Baseline at Week 60: number analyzed (Participants) | 10 | 7 | 10 | 26 | 19 | 15 | 11 | 11 | 19
  Change From Baseline at Week 60 | -1.89 (2.781) | -1.00 (1.778) | -1.63 (3.097) | -1.20 (3.371) | -2.59 (2.491) | -2.63 (3.885) | -1.17 (2.198) | -2.39 (3.217) | -2.07 (2.843)
  Change From Baseline at Week 64: number analyzed (Participants) | 10 | 7 | 10 | 26 | 19 | 16 | 12 | 13 | 19
  Change From Baseline at Week 64 | -1.19 (2.692) | -2.56 (2.525) | -0.43 (3.261) | -1.16 (2.744) | -2.05 (2.327) | -2.40 (4.271) | -1.46 (2.729) | -2.03 (4.805) | -2.38 (2.247)

27. Secondary Outcome: Change From Baseline in hsCRP Through the End of Study
Time Frame: Baseline, Weeks 4, 8, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Population: Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chronic period. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point. As pre-specified in the SAP, data is presented using the treatment sequence in the chronic period.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 14 | 14 | 46 | 27 | 30 | 26 | 26 | 29
mg/dL
  Baseline | 2.08 (2.625) | 2.41 (1.630) | 0.86 (1.942) | 1.42 (1.989) | 1.35 (1.638) | 1.22 (1.865) | 1.23 (1.687) | 1.91 (1.948) | 2.53 (1.803)
  Change From Baseline at Week 4: number analyzed (Participants) | 12 | 14 | 14 | 45 | 27 | 29 | 26 | 25 | 29
  Change From Baseline at Week 4 | -1.02 (1.888) | 0.18 (1.323) | -0.70 (1.108) | -0.43 (1.660) | -0.85 (1.585) | -0.73 (1.967) | -1.10 (1.645) | -1.40 (1.382) | -0.97 (1.656)
  Change From Baseline at Week 8: number analyzed (Participants) | 12 | 13 | 14 | 46 | 26 | 29 | 26 | 25 | 29
  Change From Baseline at Week 8 | -0.58 (2.105) | -0.22 (1.859) | -0.67 (1.957) | -0.47 (1.912) | -0.85 (2.109) | -1.14 (2.198) | -0.97 (1.980) | -1.48 (1.391) | -1.02 (1.695)
  Change From Baseline at Week 12: number analyzed (Participants) | 11 | 13 | 14 | 42 | 22 | 29 | 25 | 25 | 28
  Change From Baseline at Week 12 | -1.22 (2.248) | -0.60 (2.635) | -1.09 (2.151) | -0.66 (1.749) | -1.45 (1.768) | -1.18 (1.814) | -0.93 (2.133) | -1.50 (1.646) | -0.95 (1.646)
  Change From Baseline at Week 14: number analyzed (Participants) | 12 | 14 | 14 | 46 | 26 | 30 | 26 | 26 | 29
  Change From Baseline at Week 14 | -0.86 (2.162) | 0.08 (2.194) | -0.43 (2.529) | -0.71 (2.026) | -1.05 (2.045) | -1.10 (2.086) | -0.74 (1.750) | -1.35 (1.720) | -0.98 (1.603)
  Change From Baseline at Week 16: number analyzed (Participants) | 12 | 12 | 13 | 45 | 26 | 30 | 25 | 25 | 29
  Change From Baseline at Week 16 | -1.03 (2.061) | -0.19 (2.184) | -0.72 (2.025) | -0.56 (2.112) | -0.61 (1.931) | -1.06 (2.098) | -0.98 (2.030) | -1.50 (1.432) | -1.09 (1.783)
  Change From Baseline at Week 20: number analyzed (Participants) | 12 | 14 | 14 | 42 | 26 | 29 | 25 | 25 | 29
  Change From Baseline at Week 20 | -1.27 (1.253) | -0.98 (2.164) | -0.91 (2.855) | -0.44 (2.106) | -0.83 (2.158) | -0.52 (2.399) | -0.98 (1.957) | -0.61 (2.365) | -1.16 (1.718)
  Change From Baseline at Week 24: number analyzed (Participants) | 12 | 14 | 14 | 42 | 24 | 28 | 24 | 26 | 27
  Change From Baseline at Week 24 | -1.62 (1.786) | -1.43 (1.914) | -1.44 (1.935) | -0.53 (2.056) | -0.80 (1.811) | -0.97 (1.911) | -1.03 (1.963) | -1.48 (1.517) | -1.14 (1.639)
  Change From Baseline at Week 28: number analyzed (Participants) | 11 | 13 | 12 | 39 | 23 | 28 | 22 | 24 | 26
  Change From Baseline at Week 28 | -1.39 (1.585) | -1.00 (2.277) | -0.84 (2.000) | -0.61 (2.078) | -0.73 (2.143) | -0.76 (1.867) | -0.87 (2.125) | -1.60 (1.558) | -1.18 (1.844)
  Change From Baseline at Week 32: number analyzed (Participants) | 11 | 14 | 13 | 40 | 25 | 25 | 23 | 24 | 24
  Change From Baseline at Week 32 | -1.23 (1.930) | -0.71 (1.585) | -1.36 (1.937) | -0.58 (1.887) | -0.79 (2.136) | -0.57 (2.027) | -1.35 (1.743) | -1.15 (1.853) | -1.31 (1.988)
  Change From Baseline at Week 36: number analyzed (Participants) | 11 | 14 | 13 | 36 | 23 | 25 | 21 | 24 | 22
  Change From Baseline at Week 36 | -1.94 (2.158) | -1.21 (1.951) | -1.18 (1.032) | -0.89 (2.009) | -1.03 (2.015) | -0.95 (1.900) | -1.21 (2.006) | -1.07 (1.441) | -1.18 (1.915)
  Change From Baseline at Week40: number analyzed (Participants) | 11 | 13 | 12 | 33 | 21 | 25 | 19 | 23 | 23
  Change From Baseline at Week40 | -1.40 (2.470) | -1.03 (2.294) | -1.92 (1.184) | -0.74 (2.371) | -1.37 (2.262) | -0.84 (2.009) | -1.06 (1.992) | -1.19 (1.390) | -1.60 (1.802)
  Change From Baseline at Week 44: number analyzed (Participants) | 11 | 12 | 12 | 34 | 22 | 22 | 18 | 22 | 22
  Change From Baseline at Week 44 | -1.01 (2.243) | -1.07 (2.041) | -1.64 (1.592) | -0.99 (2.154) | -1.47 (1.876) | -0.37 (2.008) | -0.71 (1.841) | -1.03 (1.411) | -1.69 (1.423)
  Change From Baseline at Week 48: number analyzed (Participants) | 10 | 12 | 12 | 33 | 22 | 23 | 18 | 21 | 23
  Change From Baseline at Week 48 | -0.97 (1.965) | -1.06 (2.213) | -1.59 (1.530) | -0.77 (2.377) | -1.07 (1.671) | -0.78 (2.213) | -0.84 (1.802) | -1.12 (1.478) | -1.47 (1.670)
  Change From Baseline at Week 52: number analyzed (Participants) | 11 | 12 | 12 | 33 | 21 | 23 | 19 | 20 | 22
  Change From Baseline at Week 52 | -0.92 (3.093) | -0.82 (1.873) | -1.94 (1.744) | -0.94 (1.993) | -1.29 (1.756) | -1.13 (1.951) | -0.52 (1.730) | -1.22 (1.456) | -1.54 (1.863)
  Change From Baseline at Week 56: number analyzed (Participants) | 10 | 10 | 10 | 29 | 20 | 21 | 16 | 19 | 22
  Change From Baseline at Week 56 | -1.18 (2.111) | -0.96 (2.381) | -1.11 (1.681) | -0.70 (2.227) | -1.12 (2.293) | -0.71 (2.434) | -0.05 (1.966) | -0.82 (1.648) | -1.32 (2.070)
  Change From Baseline at Week 60: number analyzed (Participants) | 9 | 11 | 10 | 30 | 20 | 20 | 16 | 17 | 21
  Change From Baseline at Week 60 | -1.19 (1.259) | -0.52 (2.427) | -1.17 (2.435) | -0.64 (2.236) | -0.34 (2.332) | -0.82 (2.135) | -0.88 (2.060) | -1.71 (1.670) | -1.91 (2.213)
  Change From Baseline at Week 64: number analyzed (Participants) | 10 | 11 | 10 | 28 | 21 | 22 | 17 | 17 | 17
  Change From Baseline at Week 64 | -0.85 (1.481) | -1.03 (1.776) | -1.66 (1.908) | -0.77 (2.162) | -1.05 (1.950) | -1.22 (1.981) | -0.44 (1.778) | -1.07 (1.870) | -1.69 (2.336)

28. Secondary Outcome: Change From Baseline in Serum sTL1A Through the End of Study
Time Frame: Baseline, Weeks 4, 8, 12, 14, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 14 | 13 | 41 | 26 | 27 | 24 | 25 | 29
pg/mL
  Baseline | 6.76 (0.524) | 6.93 (0.300) | 6.89 (0.499) | 6.73 (0.503) | 6.77 (0.520) | 6.69 (0.520) | 6.83 (0.706) | 6.65 (0.467) | 6.83 (0.428)
  Change From Baseline at Week 4: number analyzed (Participants) | 12 | 14 | 13 | 39 | 25 | 27 | 24 | 24 | 29
  Change From Baseline at Week 4 | 0.09 (0.458) | -0.01 (0.349) | -0.02 (0.221) | 3.50 (1.051) | 3.73 (1.445) | 3.97 (1.218) | 4.88 (0.987) | 5.29 (0.829) | 4.65 (0.686)
  Change From Baseline at Week 8: number analyzed (Participants) | 12 | 14 | 13 | 41 | 25 | 27 | 24 | 24 | 29
  Change From Baseline at Week 8 | -0.10 (0.908) | 0.02 (0.329) | -0.10 (0.267) | 3.18 (1.331) | 3.98 (1.561) | 3.76 (1.443) | 4.87 (1.691) | 4.98 (1.434) | 4.74 (0.891)
  Change From Baseline at Week 12: number analyzed (Participants) | 11 | 12 | 13 | 39 | 23 | 27 | 23 | 25 | 29
  Change From Baseline at Week 12 | 0.14 (0.383) | -0.01 (0.329) | -0.17 (0.365) | 2.93 (1.629) | 3.84 (1.613) | 3.75 (1.471) | 4.34 (2.700) | 4.59 (1.840) | 5.03 (1.221)
  Change From Baseline at Week 14: number analyzed (Participants) | 12 | 13 | 13 | 41 | 25 | 27 | 23 | 25 | 29
  Change From Baseline at Week 14 | 0.08 (0.474) | 0.28 (1.209) | -0.23 (0.329) | 2.97 (1.598) | 3.95 (1.664) | 3.97 (1.419) | 4.37 (2.724) | 4.68 (1.872) | 5.00 (0.902)
  Change From Baseline at Week 16: number analyzed (Participants) | 11 | 12 | 13 | 39 | 24 | 26 | 23 | 25 | 29
  Change From Baseline at Week 16 | -0.05 (0.708) | 0.56 (1.384) | -0.11 (0.305) | 2.99 (1.697) | 3.55 (1.849) | 3.96 (1.406) | 4.40 (2.472) | 4.42 (2.181) | 4.66 (1.069)
  Change From Baseline at Week 20: number analyzed (Participants) | 12 | 14 | 13 | 39 | 26 | 27 | 22 | 25 | 29
  Change From Baseline at Week 20 | 4.05 (0.978) | 3.75 (1.543) | 5.19 (0.861) | 3.01 (1.710) | 3.46 (1.678) | 3.96 (1.338) | 4.12 (2.459) | 3.92 (2.248) | 4.40 (1.365)
  Change From Baseline at Week 24: number analyzed (Participants) | 12 | 13 | 13 | 37 | 22 | 25 | 22 | 24 | 27
  Change From Baseline at Week 24 | 2.94 (1.140) | 4.17 (1.415) | 5.41 (0.771) | 2.86 (1.881) | 3.57 (1.608) | 3.60 (2.046) | 3.74 (2.346) | 3.69 (2.117) | 4.33 (1.483)
  Change From Baseline at Week 28: number analyzed (Participants) | 12 | 13 | 11 | 36 | 24 | 25 | 21 | 23 | 26
  Change From Baseline at Week 28 | 3.04 (1.182) | 4.06 (1.536) | 5.67 (0.742) | 2.87 (1.992) | 3.20 (1.715) | 3.61 (2.155) | 3.55 (2.220) | 3.68 (2.141) | 4.42 (1.548)
  Change From Baseline at Week 32: number analyzed (Participants) | 11 | 14 | 12 | 36 | 23 | 23 | 21 | 23 | 24
  Change From Baseline at Week 32 | 3.29 (1.500) | 3.99 (1.497) | 5.62 (0.620) | 2.82 (1.903) | 3.09 (1.760) | 3.92 (1.535) | 3.23 (2.089) | 3.67 (2.044) | 4.39 (1.452)
  Change From Baseline at Week 36: number analyzed (Participants) | 10 | 14 | 12 | 33 | 23 | 22 | 20 | 21 | 23
  Change From Baseline at Week 36 | 3.47 (1.247) | 3.90 (1.564) | 5.55 (0.842) | 2.96 (1.813) | 3.25 (1.637) | 3.99 (1.460) | 3.12 (1.854) | 3.83 (2.020) | 4.58 (1.209)
  Change From Baseline at Week 40: number analyzed (Participants) | 11 | 13 | 11 | 32 | 21 | 23 | 18 | 22 | 24
  Change From Baseline at Week 40 | 3.56 (1.130) | 3.65 (1.865) | 5.44 (0.951) | 3.04 (1.839) | 3.02 (1.644) | 4.07 (1.582) | 2.95 (1.914) | 3.84 (2.007) | 4.42 (1.450)
  Change From Baseline at Week 44: number analyzed (Participants) | 11 | 12 | 11 | 33 | 22 | 22 | 18 | 21 | 24
  Change From Baseline at Week 44 | 3.53 (1.172) | 3.67 (1.671) | 5.34 (1.093) | 2.98 (1.762) | 2.97 (1.769) | 3.89 (1.421) | 2.90 (1.893) | 4.05 (1.823) | 4.57 (1.276)
  Change From Baseline at Week 48: number analyzed (Participants) | 11 | 12 | 11 | 32 | 22 | 22 | 17 | 20 | 23
  Change From Baseline at Week 48 | 3.47 (1.156) | 3.42 (1.682) | 5.46 (1.019) | 2.99 (1.684) | 3.01 (1.695) | 4.25 (1.438) | 3.28 (1.789) | 4.11 (1.802) | 4.61 (1.428)
  Change From Baseline at Week 52: number analyzed (Participants) | 11 | 12 | 11 | 31 | 22 | 21 | 18 | 19 | 25
  Change From Baseline at Week 52 | 3.70 (1.262) | 3.43 (1.928) | 5.43 (1.211) | 2.94 (1.668) | 3.16 (1.573) | 4.26 (1.325) | 3.10 (1.725) | 4.00 (2.021) | 4.53 (1.565)
  Change From Baseline at Week 56: number analyzed (Participants) | 10 | 12 | 9 | 28 | 19 | 21 | 16 | 18 | 23
  Change From Baseline at Week 56 | 3.83 (1.308) | 3.31 (1.961) | 5.35 (1.132) | 3.08 (1.445) | 3.00 (1.719) | 4.24 (1.510) | 3.10 (1.605) | 4.49 (1.553) | 4.74 (1.405)
  Change From Baseline at Week 60: number analyzed (Participants) | 9 | 11 | 9 | 30 | 20 | 19 | 15 | 15 | 22
  Change From Baseline at Week 60 | 3.08 (1.718) | 3.51 (1.742) | 5.07 (1.553) | 2.98 (1.710) | 3.31 (1.714) | 3.70 (1.401) | 3.26 (1.672) | 3.72 (1.928) | 4.42 (1.254)
  Change From Baseline at Week 64: number analyzed (Participants) | 10 | 11 | 8 | 27 | 21 | 20 | 15 | 17 | 21
  Change From Baseline at Week 64 | 3.31 (1.611) | 3.48 (1.919) | 4.50 (1.900) | 2.64 (2.059) | 3.30 (1.657) | 3.75 (1.383) | 2.85 (2.115) | 3.69 (2.218) | 4.39 (1.118)

29. Secondary Outcome: Chronic Period: Number of Participants With ADA and NAbs to PF-06480605
Description: as for outcome 16
Time Frame: Weeks 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60 and 64
Population: Evaluation of NAb is generally relevant only in participants who are positive for ADA. Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chronic period. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chroinc) 450 mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
Number analyzed (Participants) | 12 | 14 | 14 | 43 | 26 | 28 | 25 | 26 | 29
Participants
  ADA at Week 16: number analyzed (Participants) | 11 | 13 | 14 | 42 | 24 | 28 | 25 | 25 | 29
  ADA at Week 16 | 0 | 0 | 0 | 38 | 18 | 24 | 10 | 17 | 15
  NAb at Week 16: number analyzed (Participants) | 0 | 0 | 0 | 39 | 18 | 24 | 11 | 18 | 18
  NAb at Week 16 |  |  |  | 16 | 7 | 3 | 1 | 3 | 1
  ADA at Week 20: number analyzed (Participants) | 12 | 13 | 13 | 43 | 26 | 28 | 22 | 26 | 29
  ADA at Week 20 | 9 | 9 | 4 | 39 | 20 | 23 | 14 | 18 | 16
  NAb at Week 20: number analyzed (Participants) | 10 | 9 | 5 | 40 | 21 | 24 | 15 | 20 | 16
  NAb at Week 20 | 0 | 0 | 0 | 12 | 7 | 4 | 0 | 5 | 1
  ADA at Week 24: number analyzed (Participants) | 12 | 13 | 11 | 40 | 23 | 28 | 24 | 25 | 26
  ADA at Week 24 | 10 | 9 | 6 | 36 | 21 | 22 | 20 | 18 | 16
  NAb at Week 24: number analyzed (Participants) | 11 | 10 | 7 | 38 | 23 | 22 | 22 | 19 | 18
  NAb at Week 24 | 1 | 2 | 0 | 11 | 4 | 2 | 1 | 4 | 0
  ADA at Week 28: number analyzed (Participants) | 11 | 14 | 12 | 38 | 24 | 27 | 20 | 24 | 25
  ADA at Week 28 | 11 | 12 | 5 | 35 | 22 | 24 | 18 | 19 | 15
  NAb at Week 28: number analyzed (Participants) | 11 | 13 | 6 | 37 | 22 | 25 | 18 | 19 | 16
  NAb at Week 28 | 4 | 3 | 0 | 13 | 5 | 4 | 1 | 4 | 0
  ADA at Week 32: number analyzed (Participants) | 11 | 14 | 13 | 37 | 23 | 25 | 21 | 24 | 24
  ADA at Week 32 | 11 | 14 | 6 | 34 | 21 | 23 | 18 | 19 | 18
  NAb at Week 32: number analyzed (Participants) | 11 | 14 | 7 | 35 | 22 | 24 | 20 | 19 | 18
  NAb at Week 32 | 4 | 3 | 0 | 10 | 4 | 1 | 0 | 3 | 1
  ADA at Week 36: number analyzed (Participants) | 11 | 14 | 12 | 35 | 20 | 22 | 20 | 22 | 23
  ADA at Week 36 | 11 | 14 | 6 | 33 | 17 | 20 | 19 | 19 | 16
  NAb at Week 36: number analyzed (Participants) | 11 | 14 | 7 | 33 | 17 | 20 | 19 | 20 | 18
  NAb at Week 36 | 3 | 3 | 1 | 10 | 2 | 3 | 0 | 5 | 0
  ADA at Week 40: number analyzed (Participants) | 11 | 11 | 12 | 35 | 21 | 24 | 18 | 21 | 24
  ADA at Week 40 | 11 | 11 | 5 | 34 | 19 | 22 | 17 | 18 | 18
  NAb at Week 40: number analyzed (Participants) | 11 | 11 | 5 | 34 | 19 | 22 | 17 | 20 | 18
  NAb at Week 40 | 3 | 1 | 1 | 8 | 3 | 2 | 0 | 2 | 0
  ADA at Week 44: number analyzed (Participants) | 10 | 12 | 12 | 35 | 21 | 24 | 18 | 20 | 24
  ADA at Week 44 | 10 | 12 | 6 | 30 | 18 | 20 | 18 | 16 | 15
  NAb at Week 44: number analyzed (Participants) | 10 | 12 | 6 | 31 | 19 | 22 | 18 | 18 | 16
  NAb at Week 44 | 3 | 1 | 1 | 7 | 4 | 3 | 0 | 1 | 0
  ADA at Week 48: number analyzed (Participants) | 11 | 12 | 11 | 34 | 22 | 24 | 18 | 20 | 22
  ADA at Week 48 | 11 | 12 | 5 | 29 | 19 | 20 | 18 | 17 | 14
  NAb at Week 48: number analyzed (Participants) | 11 | 12 | 5 | 30 | 18 | 20 | 17 | 18 | 16
  NAb at Week 48 | 2 | 1 | 1 | 7 | 3 | 3 | 0 | 1 | 1
  ADA at Week 52: number analyzed (Participants) | 11 | 12 | 12 | 32 | 22 | 23 | 18 | 20 | 23
  ADA at Week 52 | 11 | 11 | 5 | 28 | 19 | 17 | 16 | 17 | 13
  NAb at Week 52: number analyzed (Participants) | 11 | 11 | 5 | 30 | 19 | 20 | 16 | 17 | 15
  NAb at Week 52 | 2 | 2 | 1 | 8 | 5 | 2 | 1 | 1 | 0
  ADA at Week 56: number analyzed (Participants) | 10 | 12 | 10 | 30 | 19 | 22 | 17 | 19 | 23
  ADA at Week 56 | 10 | 11 | 4 | 28 | 16 | 21 | 16 | 15 | 13
  NAb at Week 56: number analyzed (Participants) | 10 | 11 | 4 | 29 | 18 | 21 | 16 | 14 | 13
  NAb at Week 56 | 2 | 1 | 1 | 6 | 5 | 2 | 0 | 2 | 0
  ADA at Week 60: number analyzed (Participants) | 9 | 12 | 10 | 32 | 20 | 21 | 14 | 17 | 22
  ADA at Week 60 | 9 | 11 | 6 | 27 | 18 | 19 | 13 | 16 | 16
  NAb at Week 60: number analyzed (Participants) | 9 | 12 | 7 | 28 | 18 | 19 | 14 | 16 | 17
  NAb at Week 60 | 2 | 0 | 2 | 5 | 3 | 3 | 0 | 3 | 0
  ADA at Week 64: number analyzed (Participants) | 10 | 11 | 10 | 29 | 21 | 20 | 17 | 16 | 20
  ADA at Week 64 | 10 | 11 | 10 | 28 | 18 | 20 | 17 | 16 | 17
  NAb at Week 64: number analyzed (Participants) | 10 | 11 | 10 | 29 | 19 | 20 | 17 | 16 | 17
  NAb at Week 64 | 0 | 1 | 1 | 7 | 4 | 2 | 1 | 3 | 0

ADVERSE EVENTS:
Time Frame: Induction Period: From initiation of study treatment to either first dose in the chronic period or end of safety follow-up, whichever occurs first. (Approximately 16 weeks plus 12-week safety follow-up, if applicable.) Chronic Period: From first dose of study treatment in the chronic period to end of safety follow-up. (Approximately 40 weeks plus 12-week safety follow-up.)
Description: Safety analysis population included all participants who took at least one dose of IP during the induction period.
  Evaluable mITT population included all participants randomly assigned to IP and who took at least one dose of IP in the chronic period.
  Induction period: Results may differ from publications that used Week 14 as the end of the AE reporting timeframe.
  Chronic period: Results may differ from publications that used Week 56 as the end of the AE reporting timeframe.
Groups:
- Placebo (Induction) to PF-06480605 (Chronic) 450mg: Participants who received placebo and completed the 12-week induction period received PF-06480605, 450 mg, as a SC injection, Q4W from Week 16 to Week 52 in the chronic period.
Arm/Group | Induction Period: Placebo | Induction Period: PF-06480605 50 mg | Induction Period: PF-06480605 150 mg | Induction Period: PF-06480605 450 mg | Placebo (Induction) to PF-06480605 (Chronic) 50 mg | Placebo (Induction) to PF-06480605 (Chronic) 150 mg | Placebo (Induction) to PF-06480605 (Chronic) 450mg | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/47 | 0/62 | 0/91 | 0/12 | 0/14 | 0/14 | 0/46 | 0/27 | 0/30 | 0/26 | 0/26 | 0/29
Serious Adverse Events (participants affected / at risk) | 4/45 | 3/47 | 1/62 | 4/91 | 0/12 | 0/14 | 0/14 | 5/46 | 1/27 | 0/30 | 2/26 | 1/26 | 4/29
Other Adverse Events (participants affected / at risk) | 16/45 | 11/47 | 20/62 | 34/91 | 5/12 | 9/14 | 9/14 | 24/46 | 15/27 | 12/30 | 14/26 | 15/26 | 14/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period: Placebo (N=45) | Induction Period: PF-06480605 50 mg (N=47) | Induction Period: PF-06480605 150 mg (N=62) | Induction Period: PF-06480605 450 mg (N=91) | Placebo (Induction) to PF-06480605 (Chronic) 50 mg (N=12) | Placebo (Induction) to PF-06480605 (Chronic) 150 mg (N=14) | Placebo (Induction) to PF-06480605 (Chronic) 450mg (N=14) | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg (N=46) | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg (N=27) | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg (N=30) | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg (N=26) | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg (N=26) | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug ineffective (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period: Placebo (N=45) | Induction Period: PF-06480605 50 mg (N=47) | Induction Period: PF-06480605 150 mg (N=62) | Induction Period: PF-06480605 450 mg (N=91) | Placebo (Induction) to PF-06480605 (Chronic) 50 mg (N=12) | Placebo (Induction) to PF-06480605 (Chronic) 150 mg (N=14) | Placebo (Induction) to PF-06480605 (Chronic) 450mg (N=14) | PF-06480605 50 mg (Induction) to PF-06480605 (Chronic) 50 mg (N=46) | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 50 mg (N=27) | PF-06480605 150 mg (Induction) to PF-06480605 (Chronic) 150 mg (N=30) | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 50 mg (N=26) | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 150 mg (N=26) | PF-06480605 450 mg (Induction) to PF-06480605 (Chronic) 450 mg (N=29)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 8 (8) | 4 (4) | 2 (2) | 6 (6) | 3 (3) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (2) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 1 (5) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (9) | 2 (2) | 1 (1) | 1 (1) | 2 (4) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Chorioretinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (3) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 antibody test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 3 (3) | 4 (4) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (7) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 9 (13) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 2 (3) | 2 (3) | 1 (1)
Adnexa uteri pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04090411/Prot_002.pdf
  • Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04090411/SAP_003.pdf